CLINICAL TRIAL: NCT02905032
Title: Shared Decision Making for Stroke Prevention in Atrial Fibrillation (SDM4Afib): A Randomized Trial
Brief Title: SDM for Stroke Prevention in Atrial Fibrillation
Acronym: SDM4Afib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Park Nicollet Clinic (Other); Hennepin County Medical Center, Minneapolis (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter A. Noseworthy, M.D., M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-005409; 1R01HL131535 (NIH)
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
Keywords: Afib; Atrial fib; Shared; Decision; Making; Aid; AF
MeSH Terms: conditions — Atrial Fibrillation; Helping Behavior | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Observations in clinical encounter via video, audio or observational notes.
- Standard Care + Decision Aid (Active Comparator): Observation of clinical encounter using the decision aid via video, audio, or observational notes.
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — Observation of clinical encounter using the electronic decision aid to facilitate treatment option conversation between clinician and patient.
  Other Names: DA
  Arms: Standard Care + Decision Aid

SUMMARY:
The objective of this project is to evaluate a treatment decision aid for patients with atrial fibrillation.

DETAILED DESCRIPTION:
The goal of this study is to determine the extent to which the Anticoagulation Choice tool promotes shared decision making and its impact on anticoagulation use and adherence versus standard care in patients with nonvalvular atrial fibrillation.

ELIGIBILITY:
Clinician Inclusion Criteria:

• All clinicians (MDs, NP/PAs, PharmDs) that are responsible for the modality of Anticoagulation in eligible AF patients at participating sites, without exclusion

Patient Inclusion Criteria:

* ≥ 18 years of age
* Chronic nonvalvular atrial fibrillation deemed at high risk of thromboembolic strokes (CHA2D2-VASc Score ≥ 1, or 2 in women)
* Able to read and understand (despite cognitive, sensorial, hearing or language challenges) the informed consent document as determined by the study coordinator during consent

Patient Exclusion Criteria:

• Clinician indicates that patient is not a candidate for a discussion about anticoagulation medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Noseworthy, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Health Partners, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sivly A, Gorr HS, Gravholt D, Branda ME, Linzer M, Noseworthy P, Hargraves I, Kunneman M, Doubeni CA, Suzuki T, Brito JP, Jackson EA, Burnett B, Wambua M, Montori VM; Shared Decision-Making for Atrial Fibrillation (SDM4AFib) Trial Investigators. Enrolling people of color to evaluate a practice intervention: lessons from the shared decision-making for atrial fibrillation (SDM4AFib) trial. BMC Health Serv Res. 2022 Aug 12;22(1):1032. doi: 10.1186/s12913-022-08399-z. PMID 35962351
- [Derived] Noseworthy PA, Branda ME, Kunneman M, Hargraves IG, Sivly AL, Brito JP, Burnett B, Zeballos-Palacios C, Linzer M, Suzuki T, Lee AT, Gorr H, Jackson EA, Hess E, Brand-McCarthy SR, Shah ND, Montori VM; SDM4AFib (Shared Decision-Making for Atrial Fibrillation) Trial Investigators *. Effect of Shared Decision-Making for Stroke Prevention on Treatment Adherence and Safety Outcomes in Patients With Atrial Fibrillation: A Randomized Clinical Trial. J Am Heart Assoc. 2022 Jan 18;11(2):e023048. doi: 10.1161/JAHA.121.023048. Epub 2022 Jan 13. PMID 35023356
- [Derived] Kamath CC, Giblon R, Kunneman M, Lee AI, Branda ME, Hargraves IG, Sivly AL, Bellolio F, Jackson EA, Burnett B, Gorr H, Torres Roldan VD, Spencer-Bonilla G, Shah ND, Noseworthy PA, Montori VM, Brito JP; Shared Decision Making for Atrial Fibrillation (SDM4AFib) Trial Investigators. Cost Conversations About Anticoagulation Between Patients With Atrial Fibrillation and Their Clinicians: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116009. doi: 10.1001/jamanetworkopen.2021.16009. PMID 34255051
- [Derived] Kunneman M, Branda ME, Hargraves IG, Sivly AL, Lee AT, Gorr H, Burnett B, Suzuki T, Jackson EA, Hess E, Linzer M, Brand-McCarthy SR, Brito JP, Noseworthy PA, Montori VM; Shared Decision Making for Atrial Fibrillation (SDM4AFib) Trial Investigators. Assessment of Shared Decision-making for Stroke Prevention in Patients With Atrial Fibrillation: A Randomized Clinical Trial. JAMA Intern Med. 2020 Sep 1;180(9):1215-1224. doi: 10.1001/jamainternmed.2020.2908. PMID 32897386
- [Derived] Spencer-Bonilla G, Thota A, Organick P, Ponce OJ, Kunneman M, Giblon R, Branda ME, Sivly AL, Behnken E, May CR, Montori VM; Shared Decision Making for Atrial Fibrillation (SDM4AFib) Trial Investigators. Normalization of a conversation tool to promote shared decision making about anticoagulation in patients with atrial fibrillation within a practical randomized trial of its effectiveness: a cross-sectional study. Trials. 2020 May 12;21(1):395. doi: 10.1186/s13063-020-04305-2. PMID 32398149
- [Derived] Kunneman M, Branda ME, Noseworthy PA, Linzer M, Burnett B, Dick S, Spencer-Bonilla G, Fernandez CA, Gorr H, Wambua M, Keune S, Zeballos-Palacios C, Hargraves I, Shah ND, Montori VM. Shared decision making for stroke prevention in atrial fibrillation: study protocol for a randomized controlled trial. Trials. 2017 Sep 29;18(1):443. doi: 10.1186/s13063-017-2178-y. PMID 28962662
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Observations were in the clinical encounter via video, audio or observational notes.
- Standard Care + Decision Aid: Observation were in the clinical encounter using the decision aid via video, audio, or observational notes.
  Decision Aid: Observation of clinical encounter using the electronic decision aid to facilitate treatment option conversation between clinician and patient.
- Clinicians: Clinicians (MDs, NP/PAs, PharmDs) that are responsible for the modality of Anticoagulation in eligible atrial fibrillation patients at participating sites
Period: Overall Study
Arm/Group | Standard Care | Standard Care + Decision Aid | Clinicians
Started | 467 | 475 | 244
Completed | 459 | 463 | 244
Not Completed | 8 | 12 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 6 | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care + Decision Aid | Clinicians | Total
Number analyzed (Participants) | 459 | 463 | 244 | 1166
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Did not collect the age for 22 Clinicians
  years
    number analyzed (Participants) | 459 | 463 | 222 | 1144
    (all) | 71 (10) | 71 (11) | 42 (12) | 65 (15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Did not collect the gender for 22 Clinicians
  Participants
    number analyzed (Participants) | 459 | 463 | 222 | 1144
    Female | 191 | 172 | 112 | 475
    Male | 268 | 291 | 110 | 669
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Collected | 6 | 3 | 244 | 253
  American Indian or Alaska Native | 1 | 4 | 0 | 5
  Asian | 5 | 5 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 54 | 48 | 0 | 102
  White | 380 | 387 | 0 | 767
  Hispanic or Latino | 3 | 4 | 0 | 7
  More than one race | 8 | 10 | 0 | 18
  Unknown | 2 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 459 | 463 | 244 | 1166

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinician Satisfied Encounters
Description: The number of encounters that the clinicians were satisfied with the decision-making process. The results reported for this Outcome Measure reflect the response of the clinician for each patient. A 5 point likert scale questioning satisfaction with discussion about anticoagulation medication choice. The 5 point likert scale ranges from 1-5, with 1 being not at all satisfied and 5 being completely satisfied. Any values of 4 or 5 were considered to be satisfied.
Time Frame: 1 month
Population: Data was not analyzed nor collected for 11 subjects in Standard Care arm. Data was not analyzed nor collected for 10 subjects in Standard Care + Decision Aid arm
Measure: Number; unit: encounters
Arm/Group | Standard Care | Standard Care + Decision Aid
Number analyzed (Participants) | 448 | 453
encounters | 277 | 400

2. Primary Outcome: Number of Clinician Recommendation
Description: The number of encounters were the clinician would recommend the decision making process approach. The results reported for this Outcome Measure reflect the response of the clinician for each patient. Clinician was asked whether they would recommend the approached used to other clinician for other discussions on a 7 point Likert scale. The 7 point likert scale ranges from 1-7, with 1 being no I would strongly recommend against it and 7 being yes I would strongly recommend it. Any values of 6 or 7 were considered to be clinician would recommend.
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: encounters
Arm/Group | Standard Care | Standard Care + Decision Aid
Number analyzed (Participants) | 448 | 453
encounters | 199 | 396

3. Secondary Outcome: Number of Participants With Anticoagulant Medication Use
Description: The number of subjects who chose to start or continue receive an anticoagulant medication.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Standard Care + Decision Aid
Number analyzed (Participants) | 459 | 463
Participants | 391 | 399

4. Secondary Outcome: Patient Involvement
Description: Patient involvement in decision-making as assessed through video recordings of the encounters using the Observing Patient Involvement in Decision Making 12-item scale. The 12 items measure observed patient involvement. Each of the 12 items have possible scores that range from 0 (the behavior is not observed) to 4 (the behavior is exhibited to a very high standard). To calculate the total score for each patient, the 12 items are summed, divided by 48 (the maximum possible score), and multiplied by 100. Total score minimum is 0, maximum is 100. The higher the total score the higher the patient involvement.
Time Frame: 1 month
Population: Data was not analyzed nor collected for 48 subjects in Standard Care arm. Data was not analyzed nor collected for 44 subjects in Standard Care + Decision Aid arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Standard Care + Decision Aid
Number analyzed (Participants) | 411 | 419
score on a scale | 29.1 (13.1) | 33.0 (10.8)

5. Secondary Outcome: Encounter Duration
Description: The length of time for the subjects visit with the clinician, as measured in minutes.
Time Frame: 1 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Care | Standard Care + Decision Aid
Number analyzed (Participants) | 411 | 419
minutes | 31 (17) | 32 (16)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 months.
Arm/Group | Standard Care | Standard Care + Decision Aid | Clinicians
All-Cause Mortality (participants affected / at risk) | 19/459 | 15/463 | 0/244
Serious Adverse Events (participants affected / at risk) | 52/459 | 52/463 | 0/244
Other Adverse Events (participants affected / at risk) | 0/459 | 0/463 | 0/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=459) | Standard Care + Decision Aid (N=463) | Clinicians (N=244)
Stroke (Nervous system disorders) | 6 | 7 | NA
Major Bleeding (Blood and lymphatic system disorders) | 48 (63) | 47 (61) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT02905032/Prot_SAP_000.pdf